CLINICAL TRIAL: NCT01351636
Title: Effect of Arotinolol Hydrochloride on Cardiovascular Events in Hypertensive Haemodialysis Patients: An Open Labelled, Randomized, Multicentered, Controlled Trial
Brief Title: Effect of Arotinolol Hydrochloride on Cardiovascular Events in Hypertensive Haemodialysis Patients
Acronym: AHOCEP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sumitomo Pharma (Suzhou) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DSPC-ALM-1101
Record Dates: First submitted 2011-05-05; First posted 2011-05-11 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2015-11

CONDITIONS: Chronic Kidney Disease
Keywords: chronic kidney disease; hypertension
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hypertension | interventions — arotinolol; Almarl; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arotinolol Hydrochloride (Experimental): Antihypertensive medications plus arotinolol hydrochloride
  Interventions: Drug: Arotinolol Hydrochloride
- Non arotinolol group (Placebo Comparator): Antihypertensive medications without arotinolol hydrochloride
  Interventions: Drug: Non arotinolol group

INTERVENTIONS:
Drug: Arotinolol Hydrochloride — Antihypertensive medications plus arotinolol hydrochloride, dosage of arotinolol hydrochloride from 2.5mg bid, 2 days later increased to 5mg bid or 10mg bid, for 18 months
  Other Names: Almarl
  Arms: Arotinolol Hydrochloride
Drug: Non arotinolol group — Antihypertensive medications without arotinolol for 18 months
  Other Names: Control group
  Arms: Non arotinolol group

SUMMARY:
The purpose of this study is to ascertain whether Arotinolol Hydrochloride reduces mortality and cardiovascular events in chronic kidney disease stage 5 patients with hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18-75 years-old;
* Chronic kidney disease stage 5 with haemodialysis treatment for 2 months;
* Patients with blood pressure≥140/90 mmHg after receiving 2 or 3 antihypertensive medications for 2 weeks;
* Patients who receiving alfa or beta blockers will be washed out for 2 weeks;
* Written informed consent

Exclusion Criteria:

* Unstable angina, myocardial infarction, symptomatic or continuous arrhythmia, cardiosurgery in the last 2 months;
* Patients who taking class I antiarrhythmic drugs;
* Resting heart rate less than 60;
* Patients with systolic pressure less than 90 mmHg;
* Patients with chronic obstructive pulmonary disease and asthma;
* Patients with cerebral infarction in the last 2 weeks;
* Severe disorders of liver function;
* Allergy to the arotinolol;
* Patients who planning to have kidney transplantation in the near future;
* Pregnancy and breast-feeding;
* Malignant tumor

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2011-04 (Actual); Primary Completion 2018-10-10 (Actual); Study Completion 2018-10-10 (Actual)

PRIMARY OUTCOMES:
Composite endpoints | 18 months

SECONDARY OUTCOMES:
Changes for metabolism related index | 18 months
Blood pressure control in hypertensive haemodialysis patients | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Nan Chen, PhD, MD, Principal Investigator — Shanghai Jiaotong University Medical School Affiliated Ruijin Hospital
Locations (1):
- Nan Chen, Shanghai, Shanghai Municipality, China